CLINICAL TRIAL: NCT00922337
Title: A Prospective, Observational, Multicenter Registry To Evaluate the 'Real World' Clinical Performance of the MGuard Coronary Stent System
Brief Title: The Israeli MGuard Registry
Status: Completed | Type: Observational
Sponsor: InspireMD (Industry)
Responsible Party: Sponsor
Other Study IDs: IMD-05
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Ischemic Heart Disease; Acute Coronary Syndrome; Acute Myocardial Infarction
Keywords: distal embolization; thrombotic lesions; AMI; ACS; SVG
MeSH Terms: conditions — Myocardial Ischemia; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- MGuard: eligible patients implanted with minimum one MGuard stent
  Interventions: Device: MGuard Coronary Stent system

INTERVENTIONS:
Device: MGuard Coronary Stent system — MGuard Coronary Stent system implanted within a PCI
  Other Names: MGuard

SUMMARY:
the objective of the Israeli MGurad Registry is to evaluate the 'Real World' Clinical Performance of the InspireMD MGuard Coronary Stent System

DETAILED DESCRIPTION:
A Prospective, Observational, Multicenter Registry The primary objective of this registry is to document the safety and overall clinical performance of the MGuard Coronary Stent System in a "real world" patient population requiring stent implantation.

The secondary objective is to assess the event rate in patient subgroups with specific clinical indications and/or vessel and/or lesion characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Patient is > 18 years of age
* The patient has consented to participate by signing the "Patient Informed Consent Form"
* Patient is suitable for implantation of one or more MGuard Stent System in one or more target lesions
* Target lesion(s) are according to the Indications for Use and Israeli regulatory approval of the MGuard Stent System
* The patient is willing and able to cooperate with registry procedures and required follow up

Exclusion Criteria:

* Heavily calcified target lesions
* Target lesions with side branch bigger then 2.5mm
* Target lesions which are distal to newly stented lesion (less than 1 month).
* Women with known pregnancy
* Current medical condition with a life expectancy of less than 12 months
* Patients with medical conditions that preclude the follow-up as defined in the protocol or that otherwise limits study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an indication for coronary stent implantation according to the Israeli regulatory approval of the MGuard Coronary Stent System. All patients who receive one or more MGuard Coronary Stent System in one or more target lesions should be included.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2009-07; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Major Cardiac Adverse Events rate (MACE) | 1 month

SECONDARY OUTCOMES:
Major Cardiac Adverse Events rate (MACE) | 6 months
Lesion success rate | 1 day
Bleeding complications | 6 months
Stent thrombosis rate | 6 months
Any death | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Elad Yaacoby, Study Director — InspireMD
Locations (2):
- Israel (2):
  - Laniado Hospital, Netanya
  - Asaf Harofe Medical Center, Zrifin